CLINICAL TRIAL: NCT04452968
Title: Intermittent Fasting and Polycystic Ovarian Syndrome
Brief Title: Comparison of Intermittent Fasting and Caloric Deficit for Weight Loss in Women With Polycystic Ovarian Syndrome
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Karachi Medical and Dental College (Other)
Collaborators: Aziz Medical Center (Network)
Responsible Party: Principal Investigator, samia husain, clinical investigator, Karachi Medical and Dental College
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 33
Record Dates: First submitted 2020-06-26; First posted 2020-07-01 (Actual); Last update posted 2020-11-25 (Actual); Status verified 2020-11

CONDITIONS: Polycystic Ovarian Syndrome; Weight Loss; Intermittent Fasting
MeSH Terms: conditions — Polycystic Ovary Syndrome; Weight Loss; Intermittent Fasting | interventions — Caloric Restriction

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- intermittent fasting (Experimental): Daily caloric requirement was calculated using basal metabolic rate (BMR) calculator. All women were directed to decrease calorie intake by 500 calories.
  Women were told about timed restricted feeding. They were required to fast for 16 hours and consume their allotted calories during the remaining 8 hours.
  Interventions: Behavioral: intermittent fasting; Behavioral: Caloric restriction
- caloric restriction (Active Comparator): Daily caloric requirement was calculated using basal metabolic rate (BMR) calculator. All women were directed to decrease calorie intake by 500 calories.
  Interventions: Behavioral: Caloric restriction

INTERVENTIONS:
Behavioral: intermittent fasting — Women were required to fast for 16 hours and consume their allotted calories during the remaining 8 hours.
  Arms: intermittent fasting
Behavioral: Caloric restriction — Daily caloric requirement was calculated using basal metabolic rate (BMR) calculator. All women were directed to decrease calorie intake by 500 calories.

SUMMARY:
Time restricted feeding (TRF) has been emerging as a potential weight loss strategy that avoids major dietary changes but achieves strong effects. It also improves insulin sensitivity through increased human growth hormone. This effect helps to improve the root cause of weight gain and has additional benefits for women with PCOS.

ELIGIBILITY:
Inclusion Criteria:

* PCOS as described by Rotterdam's criteria

Exclusion Criteria:

* endocrine disorders
* diabetic
* hypertensive
* Taking medications affecting weight or energy intake/energy expenditure in the last 6 months, including weight loss medications, antipsychotic drugs or other medications as determined by the study physician;
* The body weight fluctuated more than 5% in recent 3 months.
* Liver and kidney dysfunction: renal impairment, creatinine clearance rate < 30 mL/min/1.73 m2, transaminase increased, more than three times higher than the normal limit;
* History of serious cardiovascular or cerebrovascular disease (angina, myocardial infarction or stroke) in the past 6 months;
* History of thyroid diseases;
* pregnant
* Currently participating in weight loss programs or weight change in the past 3 months (> 5% current body weight)
* Patients who cannot be followed for 16 months (due to a health situation or migration)
* Patients who are unwilling or unable to give informed consent

Ages: 20 Years to 35 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — females
Enrollment: 96 (Actual)
Dates: Start 2020-07-01 (Actual); Primary Completion 2020-10-30 (Actual); Study Completion 2020-10-30 (Actual)

PRIMARY OUTCOMES:
weight loss in kg | in 3 months

SECONDARY OUTCOMES:
decrease in body fat percentage | in 3 months
fasting plasma insulin | in 3 months
blood pressure in mm Hg | in 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Rubina Izhar, Study Chair — Aziz Medical Center
Locations (1):
- Aziz Medical Center, Karachi, Sindh, Pakistan

IPD SHARING:
Plan to Share IPD: No